CLINICAL TRIAL: NCT00674154
Title: Effect of Vitamin D Treatment in Primary Hyperparathyroidism
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHPT-20080011
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2013-10-16 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-08

CONDITIONS: Vitamin D Deficiency; Primary Hyperparathyroidism; Hypercalcemia
Keywords: Vitamin D; Primary hyperparathyroidism; hypercalcemia
MeSH Terms: conditions — Vitamin D Deficiency; Hyperparathyroidism, Primary; Hypercalcemia | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D group (Experimental): Cholecalciferol 1400 IU, 2 tablets once daily in 52 weeks
  Interventions: Drug: Cholecalciferol
- Placebo group (Placebo Comparator): Placebo, two tablets daily in 52 weeks.
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — 2800 IE daily in 52 weeks
  Other Names: vitamin D

SUMMARY:
The primary aim of the study is to assess whether 6-months of vitamin D supplements can decrease PTH compared with placebo treatment in primary hyperparathyroidism.

DETAILED DESCRIPTION:
The study investigates effects and safety of six months of vitamin D supplementation before and after surgery in primary hyperparathyroidism. Effects are assessed as changes in calcium homeostasis, bone metabolism, quality of life, and muscle strength and function.

ELIGIBILITY:
Inclusion Criteria:

* P-Ca-ion > 1,30 mmol/l
* P-PTH > 5 pmol/l
* P-OH25-vitamin D < 80 nmol/l

Exclusion Criteria:

* P-creatinin > 120 mumol/l
* usage of Etalpha, Mimpara
* Cancer
* Sarcoidosis
* malabsorption
* pancreatitis
* alcohol abuse
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Rolighed, MD, Principal Investigator; Lars Rejnmark, MD,PhD,DrMed, Study Director
Locations (1):
- Osteoporoseklinikken, Aarhus University Hospital, THG, Aarhus C, Denmark

REFERENCES:
- [Derived] Bislev LS, Wamberg L, Rolighed L, Grove-Laugesen D, Rejnmark L. Effect of Daily Vitamin D3 Supplementation on Muscle Health: An Individual Participant Meta-analysis. J Clin Endocrinol Metab. 2022 Apr 19;107(5):1317-1327. doi: 10.1210/clinem/dgac004. PMID 35018442

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We randomized 46 patients with PHPT and 25OHD-levels < 80 nmol/l to a daily supplement with 70 microgram (2800 IU) of cholecalciferol or identical placebo for 52 weeks. Accordingly, treatment was administered for 26 weeks prior to parathyroidectomy and continued for 26 weeks following surgical cure.
Pre-assignment Details: We screened 227 PHPT patients. A total of 46 patients were included.
Groups:
- Vitamin D: Cholecalciferol 1400 IE, 2 tablets once daily in 52 weeks
- Placebo: Placebo, two tablets daily in 52 weeks.
Period: Overall Study
Arm/Group | Vitamin D | Placebo
Started | 23 | 23
Completed | 20 | 20
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Did not want parathyroidectomy | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D | Placebo | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 7 | 9 | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 58 (14) | 57 (13) | 58 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  Denmark | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Decrease in Preoperative P-PTH
Description: Decrease in plasma PTH after 25 weeks of preoperative vitamin D treatment compared with the plasebo Group.
Time Frame: 25 weeks
Measure: Mean (Standard Error); unit: pmol/l
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 20 | 22
pmol/l | -2.2 (0.7) | 0.2 (1.0)

2. Secondary Outcome: Improved Muscular Function
Time Frame: One Year
Reporting Status: Not Posted

3. Secondary Outcome: Reduced Postoperative Hypocalcemia
Time Frame: Postoperative week
Reporting Status: Not Posted

4. Secondary Outcome: Increase in Quality of Life
Time Frame: One year
Reporting Status: Not Posted

5. Secondary Outcome: Increased Bone Mineral Density
Time Frame: One year
Reporting Status: Not Posted

6. Secondary Outcome: Increase in Trabecular and Cortical vBMD Measured by QCT and pQCT of Hip, Spine and Forearm
Time Frame: one year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Vitamin D | Placebo
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/22
Other Adverse Events (participants affected / at risk) | 4/20 | 6/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D (N=20) | Placebo (N=22)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) — Admission to hospital due to pain and infection from kidney stones.
Eye operation (Eye disorders) | 0 (0) | 1 (1) — Admission to hospital for operation at the eye lens.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D (N=20) | Placebo (N=22)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Upper abdominal self-limitating pain.
Steatosis hepatis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Diagnosed by chance during examination for kidney stones
Hand eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Red eczema on two fingers.
Eye infection (Eye disorders) | 1 (1) | 1 (1) — Local or bilateral eye infection.
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0) — Symptoms classified and treated as cystitis
Heamatoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Local heamatoma after tissue biopsy.
Lower leg cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Pain or cramp in one or both of the lower legs.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Respiratory infection classified and treated as pneumonia.
Voice change (Nervous system disorders) | 0 (0) | 1 (1) — Temporary voice changes after neck operation for hyperparathyroidism not classified as recurrent laryngeal nerve palsy.
Changed sense of touch (Nervous system disorders) | 0 (0) | 1 (1) — Experience of a change in the sense of touch in face, arms or legs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes